CLINICAL TRIAL: NCT02189772
Title: Randomized, Double-blind, Placebo-controlled, Multi-center, Fixed Dose Study Designed to Evaluate the Safety and Tolerability of a Single Administration of MG01CI (Metadoxine Extended Release, MDX) in Adolescents With Predominantly Inattentive Attention Deficit Hyperactivity Disorder
Brief Title: Safety and Tolerability Study of Metadoxine Extended Release (MDX) (Previously Known as MG01CI) in PI-ADHD Adolescent Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AL015
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2014-12

CONDITIONS: ADHD, Predominantly Inattentive Type
Keywords: ADHD; Inattention; MDX
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MDX (metadoxine extended release) (Experimental): Route of administration: oral
  The dose of MDX (approximately 14-22 mg/kg) will be determined by the subject's weight at the baseline visit as follows:
  * 40-49 kg 700 mg consisting of a 700 mg tablet
  * 50-64 kg 1050 mg consisting of a 700 mg tablet, a 350 mg tablet
  * 65-100 kg 1400 mg consisting of two 700 mg tablets
  Interventions: Drug: Metadoxine extended release
- placebo (Placebo Comparator): Placebo tablets will be similar in appearance (color and size) to the investigational product
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metadoxine extended release — MG01CI
  Other Names: MDX
  Arms: MDX (metadoxine extended release)
Drug: Placebo — Inactive drug
  Other Names: Sugar pill
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single administration of Metadoxine Extended Release (MDX) formulation for the treatment of adolescents diagnosed with ADHD that have predominantly inattentive symptoms. The study will also try to evaluate the efficacy of MDX and its level in the blood.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled multi-center, fixed dose, single dose study in adolescent subjects with PI-ADHD. Eligible subjects will be randomized in a 1:1 ratio to receive single administration of either MDX (approximately 14-22 mg/kg) or matching placebo.

Subjects taking a course of methylphenidate, amphetamine or atomoxetine at least two weeks prior to screening will require a 2-week wash-out (for methylphenidate, amphetamine) or a 4-week wash-out (for atomoxetine) and be requested to attend an interim screening visit.

The study will consist of three periods: a screening period of up to three weeks (and five in the case of atomoxetine washout), a 1 day treatment period, and a one-week safety follow-up period.

Overview of Study Visits Screening Period - Visit 1 (Screening/Baseline) Following signing of informed consent/assent, subjects will be screened for study eligibility. Each subject will undergo a battery of evaluations with various rating scales including Adolescent ADHD Clinical Diagnostic Scale1 (ACDS v1.2), Kiddie - Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version (K-SADS-PL), Columbia-Suicide Severity rating scale (C-SSRS), State Trait Anxiety Inventory (STAI-A and STAI-T), Beck Depression Inventory (BDI), CGI-S (Clinical Global Impression - Severity), Time-Sensitive ADHD Symptom Scale (TASS), Wechsler Intelligence Scale for Children- fourth edition (WISC-IV) sub-tests2 and Test of Variables of Attention (TOVA)3. Eligible subjects who did not require a wash-out, will be eligible for the study. In addition, the following standard assessments will be performed: assessment of inclusion/exclusion, collection of demographic data, medical history, prior medications, neurological exam, neuropathy questionnaire, physical exam, height and weight, vital signs, ECG, laboratory evaluations including hematology (complete blood count, CBC), chemistry, plasma concentration of metadoxine, urinalysis, and serum pregnancy test for women of child bearing potential. The screening visit may be conducted over multiple days. Screening visit data will be considered baseline data for statistical analysis purposes for subject requiring no washout.

Visit 1a (Interim screening visit) This visit is applicable to subjects taking medications or supplements requiring washout such as methylphenidate, amphetamine or atomoxetine at any time during the 2 weeks preceding Visit 1 (screening); these subjects will undergo a 2-week washout (for cases such as methylphenidate or amphetamine treatment) or a 4-week washout (for cases such as atomoxetine treatment) period after which they will attend an interim screening visit. Baseline TOVA, WISC-IV sub-tests1, and TASS will be performed at Visit 1a. In addition, the C-SSRS, adverse events, and concomitant medications will be recorded at this visit.

Treatment Period - Visit 2 (Day 1, visit window + 3 days) At study visit 2 (Day 1), each eligible subject will be randomized in a 1:1 allocation to receive either MG01CI or matching placebo; dose will be determined by weight at screening visit 1. Investigational product will be administered at the clinic. The WISC-IV sub-tests of Digit Span, Coding, Letter Number Sequencing, and Symbol Search will be administered. Subjects will undergo evaluations with the TOVA test 3 to 5 hours post-dose to assess their response to treatment. In addition, subjects will complete the TASS prior to administration of study drug, and 3-5 hours post-dose. At this visit, the subjects will also undergo safety assessments including urine pregnancy test (pre-dose), vital signs , neurological exam, neuropathy questionnaire, the C-SSRS and recording of adverse events (AEs) and concomitant medications. Subjects will have blood drawn for plasma concentrations of metadoxine at 1-2 hours post-dose and 3-4 hours post-dose.

Follow-Up Period - Visit 3 (Day 8, visit window ± 3 days) One week after the end of treatment, subjects will complete the TASS and will undergo safety assessments including physical exam, neurological exam, neuropathy questionnaire, vital signs, ECG, laboratory evaluations (hematology, chemistry, and urinalysis including urine pregnancy test for women of child bearing potential), the C-SSRS, and documentation of concomitant medications and AEs, if any.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent males and females, 13-17 years old, inclusive, at screening visit, with visible axillary hair.
2. Diagnosed with predominantly inattentive ADHD based on DSM V criteria for ADHD as assessed by the Adolescent ADHD Clinician Diagnostic Scale (Adol-CDS V1.2).
3. Clinical severity of at least a moderate level (Clinical Global Impression-Severity score of 4 or above).
4. STAI State score of <52, STAI Trait score of <52 and BDI score of <19.
5. Sexually active subjects of childbearing potential must agree to use an effective contraceptive throughout the study (e.g., oral contraceptives or Norplant®; a reliable double barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam]; intrauterine devices; vasectomy; or abstinence) and for at least a month after the study, and must have a negative serum pregnancy test at the Screening Visit. Females of childbearing potential are defined as women who are between menarche and 2 years post-menopause and who are not surgically sterilized. Males and Female subjects who are not sexually active, and who agree to be abstinent throughout the study, will not be required to use birth control.
6. Subject is able to attend the clinic regularly and reliably.
7. Subject is able to swallow tablets and capsules.
8. Able to understand, read, write and speak Hebrew fluently to complete study related materials.
9. Parents or legal authorized guardians (LAR), and subject, able to understand and sign written informed consent/assent to participate in the study
10. Subject and parents/LARs provide assent/consent to participate in the study. per applicable laws and regulations
11. Subject weighs ≥40 kg or ≤100 kg

Exclusion Criteria:

1. Subject has any psychiatric condition (e.g., schizophrenia or personality disorder as diagnosed by DSM-V) or clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation as determined by the investigator using medical history, physical examination, neurological examination, laboratory tests, and electrocardiograms. Common diseases such as mild hypertension, well-controlled type 2 diabetes mellitus (hemoglobin A1C <6.5%), etc, are allowed per the investigator's judgment as long as they are stable and controlled by medical therapy that is constant for at least 8 weeks before randomization and subsequently throughout the study. If there are any concerns about the suitability of the subject's medical or surgical condition, the investigator should review the subject's history with the medical monitor.
2. Subject has a known or suspected human immune deficiency virus positive status or has diseases such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.
3. Subject has a history of an allergy or sensitivity to B-complex vitamins.
4. Subject has a history of intellectual disability or a history or suspicion of autism spectrum disorder.
5. Subject has a current clinically significant Axis I diagnosis (other than ADHD) according to the K-SADS-PL or has a lifetime history of bipolar disorder or psychosis.
6. Subject has used mega-dose vitamin B6/pyridoxine during the 28 days before the Randomization Visit. Subjects will be allowed to have a 28-day washout of mega-dose vitamin B6/pyridoxine after the Screening visit. Routine multivitamin supplements will be allowed.
7. Subject has used high-dose supplements of omega-3 fatty acids ≥ 500 mg on at least 1 day (such as softgels, capsules, or fish oils; regular daily dietary consumption of fish is allowed) or folic acid supplements (other than routine multivitamin supplements) during the 2 weeks before the Randomization Visit.
8. Subject has used an investigational medication/treatment in the 30 days before the Screening Visit
9. Subject has used any medication or food supplement that the investigator or the medical monitor considers unacceptable during the 14-day period before randomization. This includes, but is not limited to, sympathomimetic agents, clonidine, guanfacine, norepinephrine reuptake inhibitors, serotonin reuptake inhibitors, sedative-hypnotics, benzodiazepines, sedating antihistamines, herbal preparations that would confound safety or efficacy assessments, and narcotics. Questions regarding the acceptability of medications and food supplements (such as melatonin) will be discussed with the medical monitor before study entry.
10. Subject has a current drug or alcohol dependence or substance abuse disorder according to DSM-V Text Revision criteria (excluding nicotine) or a history of such dependence within the last 6 months. Subject should also agree to keep their caffeine intake consistent and refrain from consuming ≥300 mg per day of caffeine (no more than three 8-ounce servings of coffee) during the study.
11. Subject has suicidality, defined as active ideation, an intent or plan, or any significant lifetime suicidal behavior (actual attempt, aborted attempt, interrupted attempt, or act or preparation towards imminently making a suicide attempt). Subjects exhibiting history (within previous 12 months) of non-suicidal self-injurious behavior will be excluded.
12. Subject has taken any prescription or non-prescription ADHD medications during the 14 days before the randomization visit or 28 days in the case of atomoxetine..
13. Subject is significantly visually impaired to an extent that is not able to be corrected by prescription glasses or contact lenses
14. Subject is closely related to the sponsor, investigator, or study staff. Eligibility of subjects with any relationship to the sponsor, investigator, or study staff will be discussed with the medical monitor before study entry.
15. Subject has any condition that, in the principal investigator's opinion, would place the subject at risk or influence the conduct of the study or interpretation of results, including (but not limited to) abnormally low intellectual capacity as judged by the investigator.
16. Subject cannot fully comprehend the implications of the protocol, cannot comply with its requirements, or is incapable of following the study schedule for any reason.
17. Subject is pregnant, lactating, or using an inadequate contraceptive method.
18. Subject is not currently participating in other clinical trials.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 6 weeks
  Frequency of treatment emergent adverse events (AEs). Frequency of subjects who withdrew early from the study due to AE.

SECONDARY OUTCOMES:
Efficacy | Up to 5 weeks
  Change in TOVA 8 API from Baseline to 3-5 hours post-dose for all subjects and for subjects who have an abnormal TOVA 8 API at baseline (score <0). Change in TOVA sub-scores1 from Baseline to 3 -5 hours post-dose for all subjects and for subjects who have an abnormal TOVA 8 API at baseline (score<0).
  TOVA Response Rates: Change in TOVA 8 API from abnormal (ADHD score below zero, sub-scores below 85) to normal value post-dose. Improvement of 0.8 points in TOVA 8 API or 8 points in any sub-score for all subjects and for those subjects who have an abnormal TOVA 8 API at baseline (score<0).
  Change in each of WISC-IV subtests (Digit Span, Coding, Letter Number Sequencing, and Symbol Search) from Baseline to post-dose. Change in Working memory and Processing Speed from Baseline (derived from subtests)
PK | Up to 5 weeks
  Blood samples for baseline plasma concentration of metadoxine will be collected at Screening. On study visit 2 (Day 1), subjects will have another PK blood sample at 1-2 hours and 3-4 hours post-dose. The PK samples will be sent to the bioanalysis laboratory for assay.

OTHER OUTCOMES:
Exploratory endpoint | Up to 5 weeks
  Change in TASS score from Baseline to 3-5 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Iris Manor, MD, Principal Investigator — ADHD Unit, Geha Medical Center, Petah Tikva, Israel
Locations (6):
- Israel (6):
  - Rambam Medical Center, Haifa, Israel
  - Hadassah-Hebrew University Medical Center,, Jerusalem, Israel
  - Geha Medical Centre, Petah Tikva, Israel
  - The Chaim Sheba medical center, Tel Hashomer, Ramat Gan, Israel
  - Assaf Harofeh MC, Zrifin, Israel
  - Shalvata Mental Health Center, Hod HaSharon